CLINICAL TRIAL: NCT01533415
Title: The Efficacy of Cranial-electrotherapy Stimulation (CES) Using Alpha-Stim Technology in The Treatment of Anxiety Disorders
Brief Title: Use of Alpha-Stim Cranial-electrotherapy Stimulation (CES) in the Treatment of Anxiety
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyndhurst Counseling Center (Other)
Collaborators: Liberty University (Other)
Responsible Party: Principal Investigator, Tim Barclay, Asst. Professor, Wyndhurst Counseling Center
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1241.020712
Record Dates: First submitted 2012-02-11; First posted 2012-02-15 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Anxiety
Keywords: Anxiety; Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders | interventions — Patient Health Questionnaire

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active CES treatment (Active Comparator): Out of the total population of 150 participants,75 of them will be assigned to the active treatment group. Because this is a double-blind study it is unknown which members will belong to this group until completion of the study.
  Interventions: Device: CES treatment using Alpha-Stim technology
- Sham CES treatment (Sham Comparator): Of the 150 participants in this study, half of them will be assigned to the sham treatment group. Because this is a double-blind study, it is unknown which members will be assigned to this group until the completion of the study.
  Interventions: Device: Shame CES Treatment

INTERVENTIONS:
Device: CES treatment using Alpha-Stim technology — Treatment involves the passage of micro current levels of electrical stimulation across the head via electrodes placed bilaterally on the ears. The current used in this device is no stronger than the current that naturally occurs in the human body. Treatment is delivered using a current equal to 0.5 Hz for a period of 60 mins. Treatment will be self-administered on a daily basis 5-7 days per week.The manufacturer of the device, Electro medical Products, Inc. will provide the devices for the study. They will alter the functional devices to deliver treatment at a therapeutic level of <1 mA. The current cannot be altered by the participant. Participants will be required to log the date, time, and duration of treatment. The logs will be provided by the PI and will be collected weekly. Participants will also be required to complete the Hamilton Anxiety Rating Scale (HAM-A) and the Hamilton Depression Rating Scale 17 (HAM-D17) at baseline and at weeks 1, 3, and 5.
  Other Names: Alpha-Stim; CES; Anxiety
  Arms: Active CES treatment
Device: Shame CES Treatment — Treatment will be self-administered on a daily basis 5-7 days per week.The manufacturer of the device, Electro medical Products, Inc. will provide the devices for the study. They will alter the devices so they cannot emit an electrical current. The ability for the device to emit a current cannot be altered by the participant. Participants will be required to log the date, time, and duration of treatment. The logs will be provided by the PI and will be collected weekly. Participants will also be required to complete the Hamilton Anxiety Rating Scale (HAM-A) and the Hamilton Depression Rating Scale 17 (HAM-D17) at baseline and at weeks 1, 3, and 5.
  Other Names: Alpha-Stim; CES; Anxiety
  Arms: Sham CES treatment

SUMMARY:
Is CES effective in the treatment of anxiety when accounting for any comorbid conditions and or current treatments including medication and psychotherapy.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the efficacy of Alpha-Stim technology in the treatment of anxiety by using a double-blind clinical trial over a period of five weeks. Cranial-electrotherapy stimulation (CES) is a noninvasive procedure that has been used for decades in the United States to treat anxiety, depression, and insomnia. Although many studies on CES have been published in previous decades, most have used relatively small samples using various frequencies and links of treatment. Given the positive results of the many general studies that have been performed to date, this study seeks to add to the current literature by addressing previous criticisms using a large sample size (n=150)and using participants that represent more than a single type of anxiety along with comorbidity. Such a population is believed to better represent typical treatment complications.

Participants will be recruited via advertisements in a local newspaper and posting of flyers around a local university campus. Participants will be screened through an intake process using the Structured Clinical Interview for Axis I Disorders (SCID-I) to confirm a diagnosis of an anxiety disorder. Comorbid conditions are acceptable, however, an anxiety disorder must be the primary diagnosis. As part of the intake process, participants will complete the Hamilton Anxiety Rating Scale (HAM-A)and the Hamilton Depression Rating Scale (HAM-D17) to establish a baseline. These instruments will serve as the primary efficacy measures. In order to participate, HAM-A scores must equal to or greater than 18 (Moderate Anxiety). Depression will be monitored using The HAM-D17 as depression is a commonly occurring condition with anxiety and the HAM-D17 is also sensitive to anxiety. Current treatment with medications are also acceptable provided there will be no changes in dosage or type during the study. See Inclusions and Exclusions for further information. All participants will pay a fee of $30 to enter the study to cover administration costs and as a way to measure placebo effect. Participants will be assigned a device to take home and self-administer treatment 5-7 days a week. Participants will be required to log their treatment times and dates with logs provided by the researcher. The student population will not be given a take home device but will receive treatment at the Graduate Assistant's Office or Student Care Office.

Electromedical Products International, Inc. has agreed to supply the devices needed to carry out the research to include conductance solution, felt tabs, and batteries. Half of the devices will be set by the manufacturer to deliver treatment at 0.5 Hz and at the lowest therapeutic setting. The remaining devices will be shame and not deliver any therapeutic benefit. The devices will not be able to be altered by the participant.

Participants will meet with the PI or research assistant to complete the HAM-A and HAM-D17 at weeks 1, 3, and 5 at a designated location either in the researchers private practice office or university lab location. Adverse treatment reactions will also be noted. Treatment logs will also be collected at these points. At weeks 1 and 3, participants will be given fresh batteries, conductance solution, and felt tabs as needed. At the completion of the study, participants found to be in the shame treatment group will be offered the normal course of treatment. Participants not wanting to continue the study or do not wish to follow through with normal treatment after being in the shame group will be refunded their fee.

The hypothesis this study seeks to address is:

H°: There is no difference between sham treatment and active CES on level of anxiety as compared to scores on the HAM-A and HAM-D17.

H¹ : The active CES treatment group has significantly lower anxiety scores on the HAM-A and HAM-D17 than the sham group at the endpoint of the study.

Statistical analysis will compare baselines scores (week 1) to midpoint scores (week, 3), and scores at the endpoint of the study (week 5). Response to treatment will be defined as an improvement of 30% or greater on the HAM-A and HAM-D17 at the endpoint of the study. The impact of prescription medication as a confounding variable in relation to the effect of CES on anxiety and depression will also be examined. Data analysis will consist of a repeated measures design that will likely use a general linear model in SPSS and hierarchical linear and quadratic growth models to assess individual change. The reason for this approach is that hierarchical analysis of individual change is advantageous when there are multiple repeated measure data patterns because it affords the research an opportunity to combine into a single analysis (Raudenbush & Byrk, 2002). We will estimate both the individual growth and mean growth for each point in the time series. Cross-validation of quadratic will occur via the estimation of a piecewise linear growth models to assess whether growth is more variable for one period over another during the study time frame.

Optimal design software has been used to make a preliminary determination that 100 or more participants in a randomized quadratic growth individual change model will achieve a power of .80 to .95 for a study expecting an effect size of between 0.6 to .80, respectively (0.62 is premised upon meta-analysis for CES undertaken by Klawansky, et al., 1995 and .8 is considered a large effect by Cohen, 1988). We will employ power analysis again once sample size is confirmed following recruitment of participants and expect upwards of 150 or more participants. Missing data will be explained using an intent-to-treat analysis whereby we employ redundant analysis procedures (i.e., survival analysis) to understand and context the true treatment effect.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female outpatients age 18 to 65 years.
* The subject meets DSM-IV criteria for an anxiety disorder.
* Participants with comorbidity must carry an anxiety disorder as a primary diagnosis.
* Written informed consent must be obtained from the subject prior to study participation.
* The subject is in good medical health or with chronic medical conditions which are currently stable.
* No current abuse of alcohol or other substance.
* The subject has a total score greater than 15 on the Beck Anxiety Inventory and a score greater than 45 on the Zung Self Report Anxiety Scale.

Exclusion Criteria:

* The subject meets DSM-IV criteria for an Axis I diagnosis (other than an Anxiety Disorder) as the primary diagnosis (i.e., schizophrenia, mood disorder, psychosis, anorexia nervosa).
* The subject is clinically judged by the investigator to be at risk for suicide or is acutely suicidal.
* The subject is clinically judged by the investigator to be at risk for homicide or is acutely homicidal.
* The subject has a psychiatric condition that would require inpatient, or partial psychiatric hospitalization.
* Seizure disorders.
* Significant history of medical disease (i.e. cardiovascular, hepatic (e.g. cirrhosis, hepatitis B or C) renal, gynecological, musculoskeletal, neurological, gastrointestinal, metabolic, hematological, endocrine, cancer with a metastatic potential or progressive neurological disorders) which could impair reliable participation in the trial or necessitate the use of medication not allowed by this protocol.
* Use of a pacemaker.
* The subject is pregnant, planning to become pregnant, or nursing. If a subject becomes pregnant, she will be discontinued immediately and followed appropriately.
* Current psychotherapeutic treatment except for treatment with Specific Reuptake Inhibitor (SSRIs) medications which include: Fluoxetine (Prozac), Paroxetine (Paxil), Sertraline (Zoloft), Luvox (Fluvoxamine), Citalopram. Potential subjects may remain on their medications provided that he or she has been on a stable dose prior to entering this study; the dose and type of medication remains stable throughout the remainder of this study; and it can be determined that this medication is not exacerbating the anxiety symptoms.
* History of poor compliance or in the Investigator's judgment patients any subject whose treatment as an outpatient would be clinically contraindicated
* The subject has attempted suicide one or more times within the past twelve months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Anxiety symptoms as reported on the Hamilton Anxiety Rating Scale | Change from Baseline in Hamilton Anxiety Rating Scale scores assessed at different points, e.g., Week 1, Week 3, and Week 5.
  The HAM-A was one of the first rating scales developed to measure the severity of anxiety symptoms, and is still widely used today in both clinical and research settings. The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Scores range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Depression symptoms as reported on the Hamilton Depression Rating Scale 17 | Change from Baseline in Hamilton Depression Rating Scale 17 scores assessed at different points, e.g., Week 1, Week 3, and Week 5.
  The Hamilton Depression Scale is a test measuring the severity of depressive symptoms in individuals. It is often used as an outcome measure of depression in research. In the 17-item version, nine of the items are scored on a five-point scale, ranging from zero to four. The remaining eight items are scored on a three-point scale. For the 17-item version, scores can range from 0 to 54. 0 and 6 indicate a normal person with regard to depression, scores between 7 and 17 indicate mild depression, scores between 18 and 24 indicate moderate depression, and scores over 24 indicate severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Tim H Barclay, Ph.D., Principal Investigator — Liberty University
Locations (2):
- United States (2):
  - Liberty Univeristy Student Care and Grad.Assist Office, Lynchburg, Virginia
  - Wyndhurst Counseling Center, Lynchburg, Virginia

REFERENCES:
- [Background] Klawansky S, Yeung A, Berkey C, Shah N, Phan H, Chalmers TC. Meta-analysis of randomized controlled trials of cranial electrostimulation. Efficacy in treating selected psychological and physiological conditions. J Nerv Ment Dis. 1995 Jul;183(7):478-84. doi: 10.1097/00005053-199507000-00010. PMID 7623022
- [Derived] Barclay TH, Barclay RD. A clinical trial of cranial electrotherapy stimulation for anxiety and comorbid depression. J Affect Disord. 2014 Aug;164:171-7. doi: 10.1016/j.jad.2014.04.029. Epub 2014 Apr 21. PMID 24856571